CLINICAL TRIAL: NCT00898833
Title: Laboratory Studies in Hormone Refractory Prostate Cancer - A Companion Study to CALGB 9480 and 9583
Brief Title: Plasma and Urine Samples From Patients With Hormone-Refractory Prostate Cancer Enrolled on Clinical Trials CALGB-9480 or CALGB-9583
Status: Terminated | Type: Observational
Why Stopped: The proposed work could not be completed.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-150201; CALGB-150201; CDR0000321397 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage III prostate cancer; stage IV prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Plasma, serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Previously collected plasma and urine samples are analyzed for VEGF via ELISA, plasma samples are analyzed for CgA and IL-6 via ELISA, hK2 via immunometric assay, plasma samples are analyzed for PSA via Tandem-R PSA kit, plasma samples are analyzed for TNF-alpha, sTNF-R1, and IL-8 via quantikine IL-8 immunoassay.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and urine from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This laboratory study is measuring plasma and urine biomarkers in patients with advanced prostate cancer that did not respond to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Correlate plasma and urine vascular endothelial growth factor (VEGF) levels with survival duration in patients with advanced hormone-refractory adenocarcinoma of the prostate previously enrolled on CALGB-9480.
* Determine whether plasma chromogranin A (CgA) and plasma interleukin-6 (IL-6) levels predict survival duration in these patients.
* Determine whether plasma human Kallikrein 2 (hK2) levels are prognostic for overall survival of these patients.

Secondary

* Determine the prognostic significance of plasma and urine VEGF levels, plasma CgA levels, plasma IL-6 levels, and plasma hK2 levels in relation to overall survival of these patients.
* Correlate plasma VEGF levels with urine VEGF levels in these patients.
* Correlate plasma CgA levels with previously measured serum prostate-specific antigen (PSA) and plasma VEGF levels in these patients.
* Correlate plasma hK2 levels with PSA changes after treatment with suramin to determine if hK2 may have predictive value, independent or additive to measures of disease response in these patients.
* Correlate plasma hK2 levels with PSA levels in these patients.

OUTLINE: Plasma from patients is collected for measurement of the following biomarkers: vascular endothelial growth factor (VEGF), chromogranin A, interleukin-6, and human Kallikrein 2. Urine is collected for VEGF measurement.

ELIGIBILITY:
* Registration to CALGB 9480 or 9583
* Samples collected and shipped appropriately
* Institutional Review Board (IRB) review and approval at the institution where the laboratory work will be performed is required

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hormone refractory prostate cancer enrolled on CALGB-9480 or 9583
Sampling Method: Non-Probability Sample
Enrollment: 868 (Estimated)
Dates: Start 2003-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Confirmation of plasma VEGF levels inversely correlate with survival time | Up to 3 years
Confirmation of urine VEGF levels inversely correlate with survival time | Up to 3 years
CgA levels in predicting survival time | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ellen Taplin, MD, Study Chair — Dana-Farber Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States